CLINICAL TRIAL: NCT01647893
Title: A Phase 1 Clinical Study, Randomized, Double-blind, Placebo-controlled, Single-dose, Dose Escalation Study of the Safety and Pharmacokinetic/Pharmacodynamic Profiles of CTB-001 Intravenously Administered in Healthy Male Subjects
Brief Title: Phase 1 Single Dose Escalation Study of CTB-001
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HLB Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CTB-001
Record Dates: First submitted 2012-07-17; First posted 2012-07-24 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
MeSH Terms: interventions — bivalirudin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- CTB-001 or placebo(mannitol) 0.375mg/kg, single-dose (Experimental)
  Interventions: Drug: CTB-001
- CTB-001 or placebo(mannitol) 0.75mg/kg, single-dose (Experimental)
  Interventions: Drug: CTB-001
- CTB-001 or placebo(mannitol) 1.5mg/kg, single-dose (Experimental)
  Interventions: Drug: CTB-001
- CTB-001 or placebo(mannitol) 0.75mg/kg, and dose escalation (Experimental)
  Interventions: Drug: CTB-001

INTERVENTIONS:
Drug: CTB-001 — IV bolus or IV infusion

SUMMARY:
A Phase 1 Clinical Study, Randomized, Double-blind, Placebo-controlled, Single-dose, Dose Escalation Study of the Safety and Pharmacokinetic/Pharmacodynamic Profiles of CTB-001 Intravenously Administered in Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 20 to 40 years at screening.
* Be able to understand the objective, method of the study, the characteristics of investigational drug, and comply with the requirement of the study. Subject must provide written informed consent prior to study participation.

Exclusion Criteria:

* History or presence of liver, kidney, or nervous system disease, respiratory disorders, endocrinological disorders, hemato-oncologic, cardiovascular or psychiatric or cognitive disorders.
* History of gastrointestinal disorders (bleeding, ulceration, hemorrhoids, piles) or disorders of absorption, distribution, metabolism, excretion.
* History of known hypersensitivity to drugs including CTB-001

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Safety | Up to 7 hours
  Summary statistics for SAD parts will be prepared for measured values and changes from baseline values for each dose group. Placebo subjects will serve as the control. Summaries of treatment-emergent and clinically important abnormalities in ECG, physical examination, vital signs, and laboratory (clinical chemistry, hematology, coagulation, urinalysis) data will be provided. The incidence of adverse events(AEs) will be tabulated and compared across dose group in the SAD parts.

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea